CLINICAL TRIAL: NCT02540954
Title: An Open-label, Randomized, Active-controlled, Parallel-group, Phase-3b Study of the Efficacy, Safety, and Tolerability of 2 mg Aflibercept Administered by Intravitreal Injections Using Two Different Treatment Regimens to Subjects With Neovascular Age-related Macular Degeneration (nAMD).
Brief Title: Efficacy and Safety of Two Different Aflibercept Regimens in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16598; 2013-000120-33 (EudraCT Number)
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Macular Degeneration
Keywords: Age-related macular degeneration (AMD); Eylea treatment; Treat and Extend; Intravitreal
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aflibercept extended dosing (Experimental): Aflibercept was administered 2mg per injection intravitreal (IVT) in the study eye in Aflibercept extended dosing. Flexible dosing interval is ≥ 8 weeks (no upper limit) based on visual and anatomic outcomes as judged by the investigator. When/if visual and anatomical outcomes indicated that the disease had re-activated, the treatment interval reverted to the last treatment interval in which the disease was inactive (ie, no signs of exudation were observed).
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Aflibercept 2Q8 (2 mg aflibercept administered every 8 weeks) (Active Comparator): Aflibercept was administered 2mg per injection IVT in the study eye in Aflibercept 2Q8. Fixed dosing interval is 8 weeks (±3 days), modification of the treatment interval was not allowed.
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — A dose of 2 mg aflibercept injected intravitreally

SUMMARY:
To compare the efficacy of 2 mg aflibercept administered by two different intravitreal (IVT) treatment regimens to subjects with neovascular age-related macular degeneration (nAMD)

DETAILED DESCRIPTION:
330 Patients who have completed at least one year of treatment with aflibercept will be randomized to two different aflibercept regimens and followed for 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The following criteria must have been met at the initial start of aflibercept treatment (i.e. start of aflibercept treatment at least 1 year before this study):

  * Subject had primary subfoveal choroidal neovascularization (CNV) lesions secondary to nAMD, including juxtafoveal lesions that affect the fovea, as evidenced by fluorescein angiography/photography (FA/FP) of the study eye within 3 weeks before the initiation of aflibercept treatment.
  * The area of CNV occupied at least 50% of the total lesion within 3 weeks before the initiation of aflibercept treatment.
  * Documented best-corrected visual acuity (BCVA) was 20/40 to 20/320 (letter score of 73 to 25) in the study eye at the initiation of treatment.
* Men and women >= 51 years of age
* The subject's history of aflibercept treatment meets ALL of the following:

  * Treatment in the study eye was initiated with three monthly (-1 week/+2 weeks) doses of 2 mg aflibercept and improvements of visual and anatomic outcomes were observed
  * Following the above initiation phase, the intervals between treatments were between 6 weeks and 12 weeks

Exclusion Criteria:

- Any prior or concomitant therapy with an investigational or approved agent to treat neovascular AMD in the study eye other than aflibercept.

* Total lesion size > 12 disc areas (30.5 mm2, including blood, scars and neovascularization) as assessed by fluorescein angiography (FA) in the study eye
* Subretinal hemorrhage that was:

  1. 50% or more of the total lesion area, or
  2. if the blood was under the fovea, and
  3. the blood under the fovea was 1 or more disc areas in size in the study eye.
* Scar or fibrosis making up more than 50% of the total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* Causes of CNV other than AMD in the study eye.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- Vienna, Austria
- Canada (2):
  - Toronto, Ontario
  - Clinique medicale de l'oeil de l'Estrie, Sherbrooke, Quebec
- Czechia (3):
  - Hradec Králové
  - Pilsen
  - Prague
- France (6):
  - Paris, Cedex 12
  - Bordeaux
  - Dijon
  - Lyon
  - Nice
  - Paris
- Germany (9):
  - Würzburg, Bavaria
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Düsseldorf, North Rhine-Westphalia
  - Leipzig, Saxony
  - Berlin
  - Hamburg
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Italy (9):
  - Rome, Lazio
  - Genoa, Liguria
  - Brescia, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
  - Catania, Sicily
  - Pisa, Tuscany
  - Verona, Veneto
  - Parma
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (2):
  - Gdansk
  - Olsztyn
- Portugal (4):
  - Coimbra
  - Leiria
  - Lisbon
  - Porto
- Slovakia (2):
  - Bratislava
  - Nitra
- Spain (3):
  - L'Hospitalet de Llobregat, Barcelona
  - Barcelona
  - Valencia
- Switzerland (2):
  - Bern
  - Geneva
- United Kingdom (14):
  - Southampton, Hampshire
  - Liverpool, Merseyside
  - Great Yarmouth, Norfolk
  - Middlesbrough, North Yorkshire
  - Pont-y-clun, Rhondda, Cynon, Taff
  - Guildford, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Sunderland, Tyne and Wear
  - Rugby, Warwickshire
  - Wakefield, West Yorkshire
  - Hull, York
  - Colchester
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Kodjikian L, Arias Barquet L, Papp A, Kertes PJ, Midena E, Ernest J, Silva R, Schmelter T, Niesen T, Leal S. Intravitreal Aflibercept for Neovascular Age-Related Macular Degeneration Beyond One Year of Treatment: AZURE, a Randomized Trial of Treat-and-Extend vs. Fixed Dosing. Adv Ther. 2024 Mar;41(3):1010-1024. doi: 10.1007/s12325-023-02719-3. Epub 2024 Jan 6. PMID 38183525
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 76 centers in 14 countries or regions, between 29-SEP-2015 (first participant first visit) and 04-JUN-2020 (last participant last visit)
Pre-assignment Details: At baseline, 336 participants were randomized to one of 2 treatment groups; 168 participants were randomized to the extended-dosing group and 168 participants were randomized to the 2Q8 (2 mg aflibercept administered every 8 weeks) group.
Period: Overall Study
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Started (Randomized) | 168 | 168
Treated | 167 | 168
Post-baseline BCVA Assessment | 165 (FAS) | 167 (FAS)
Completed | 149 (Completed treatment) | 154 (Completed treatment)
Not Completed | 19 | 14
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Death | 0 | 3
Not completed — Treatment failure | 1 | 0
Not completed — Other reason | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): included all participants who received any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks) | Total
Number analyzed (Participants) | 167 | 168 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (8.3) | 74.7 (7.0) | 75.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 108 | 215
  Male | 60 | 60 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 136 | 128 | 264
  Unknown or Not Reported | 31 | 40 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 139 | 132 | 271
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 36 | 64
Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual [Mean (Standard Deviation); unit: Letters read correctly] — Visual function was assessed with the procedure from the ETDRS adapted for the Age Related Eye Disease Study using charts with 70 letters at a starting distance of 4 meters. Charts are organized in 14 lines of decreasing size with 5 letters each. Participants reading up to 19 letters at 4 meters were tested at 1 meter to read the first 6 lines. The score equals the sum of letters read at 1 meter and 4 meters. If more than 19 letters are read at 4 meters the score equals the number of letters read plus 30. The score range is 0 to 100, and a higher score represents better visual function. Population: The Full Analysis Set included all randomized subjects who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
  Letters read correctly
    number analyzed (Participants) | 165 | 167 | 332
    (all) | 69.0 (12.1) | 70.1 (10.9) | 69.6 (11.5)
Central retinal thickness (CRT) in the study eye [Mean (Standard Deviation); unit: μm] — Retinal characteristic was evaluated using Optical coherence tomography (OCT). Population: The Full Analysis Set included all randomized subjects who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
  μm
    number analyzed (Participants) | 165 | 167 | 332
    (all) | 257.3 (67.8) | 264.4 (59.7) | 260.9 (63.8)
Choroidal neovascularization (CNV) area in the study eye [Mean (Standard Deviation); unit: mm*2] — Choroidal neovascularization measured by optical coherence tomography (OCT). Population: The Full Analysis Set included all randomized subjects who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
  mm*2
    number analyzed (Participants) | 165 | 167 | 332
    (all) | 4.695 (4.043) | 5.060 (4.105) | 4.875 (4.070)
Total score for National Eye Institute 25-Item Visual Function [Mean (Standard Deviation); unit: Score on a scale] — National Eye Institute 25-Item Visual Function Questionnaire (NEI VFQ-25) total score ranges from 0 to 100, where 100 represents the best possible score and 0 represents the worst. Population: The Full Analysis Set included all randomized subjects who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
  Score on a scale
    number analyzed (Participants) | 165 | 167 | 332
    (all) | 72.889 (18.414) | 75.757 (15.495) | 74.340 (17.034)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) Letter Score for the Study Eye
Description: Visual function was assessed with the procedure from the ETDRS adapted for the Age Related Eye Disease Study using charts with 70 letters at a starting distance of 4 meters. Charts are organized in 14 lines of decreasing size with 5 letters each. Participants reading up to 19 letters at 4 meters were tested at 1 meter to read the first 6 lines. The score equals the sum of letters read at 1 meter and 4 meters. If more than 19 letters are read at 4 meters the score equals the number of letters read plus 30. The score range is 0 to 100, and a higher score represents better visual function.
Time Frame: From baseline to Week 52
Population: The outcome measure was analyzed based on full analysis set (FAS). The FAS included all randomized participants who received any study drug and had a baseline BCVA assessment and at least one post-baseline BCVA assessment.
Measure: Mean (Standard Deviation); unit: Letters read correctly
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
Letters read correctly | -0.3 (7.5) | -0.5 (8.4)
Statistical Analysis 1: Comparison: Aflibercept Extended Dosing vs Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks); Test type: Non-Inferiority — Non-inferiority margin is 5 letters; p < 0.0001, ANCOVA; Least squares mean difference = 0.22, 95% CI 2-sided [-1.51 to 1.96]

2. Secondary Outcome: Percentage of Participants Maintaining Vision in the Study Eye
Description: A participant was classified as maintaining vision if the participant had lost fewer than 15 letters in the ETDRS letter score compared to baseline.
Time Frame: At week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
Percentage of participants | 95.2 | 94.0
Statistical Analysis 1: Comparison: Aflibercept Extended Dosing vs Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks); Test type: Non-Inferiority — Non inferiority margin is 7%; Treatment difference in % = 1.1, 95% CI 2-sided [-3.7 to 6.0]

3. Secondary Outcome: Percentage of Participants Who Gained From Baseline 5 or More Letters in the Study Eye
Time Frame: At week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
Percentage of participants | 24.2 | 21.0

4. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: Retinal characteristic was evaluated using Optical coherence tomography (OCT).
Time Frame: From baseline to week 52
Population: The outcome measure was analyzed based on full analysis set (FAS) with number of participants evaluable for this specific end point.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
μm | -24.4 (55.2) | -33.4 (47.1)

5. Secondary Outcome: Mean Change From Baseline in Choroidal Neovascularization (CNV) Area in the Study Eye
Description: Choroidal neovascularization measured by optical coherence tomography (OCT).
Time Frame: From baseline to week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm*2
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
mm*2 | 0.274 (2.723) | 0.204 (2.813)

6. Secondary Outcome: Percentage of Participants Who Lost From Baseline 30 or More Letters in the Study Eye
Time Frame: At week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
Percentage of participants | 0 | 0.6

7. Secondary Outcome: Mean Change From Baseline in Total Score for National Eye Institute 25-Item Visual Function (NEI VFQ-25) Questionnaire
Description: National Eye Institute 25-Item Visual Function Questionnaire (NEI VFQ-25) total score ranges from 0 to 100, where 100 represents the best possible score and 0 represents the worst.
Time Frame: From baseline to week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 165 | 167
Score on a scale | 0.186 (9.601) | -1.694 (10.328)
Statistical Analysis 1: Comparison: Aflibercept Extended Dosing vs Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks); Test type: Other; Mean Difference (Final Values) = -1.880, 95% CI 2-sided [-4.152 to 0.392]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Time Frame: Started after the first application of aflibercept in the study and less than or equal to 30 days after the last dose of study drug over approximately 1.5 years
Population: Number of participants with TEAE was analyzed based on safety analysis set (SAF) with number of participants evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
Number analyzed (Participants) | 167 | 168
Participants
  Any TEAE | 130 | 124
  Any serious TEAE | 26 | 23

ADVERSE EVENTS:
Time Frame: From after the first application of aflibercept in the study to 30 days after the last dose of study drug over approximately 1.5 years.
Arm/Group | Aflibercept Extended Dosing | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/167 | 3/168
Serious Adverse Events (participants affected / at risk) | 26/167 | 23/168
Other Adverse Events (participants affected / at risk) | 60/167 | 70/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept Extended Dosing (N=167) | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks) (N=168)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Retinal haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oesophageal prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept Extended Dosing (N=167) | Aflibercept 2Q8 (2 mg Aflibercept Administered Every 8 Weeks) (N=168)
Cataract (Eye disorders) | 17 (22) | 19 (27)
Visual acuity reduced (Eye disorders) | 14 (18) | 4 (6)
Choroidal neovascularisation (Eye disorders) | 9 (10) | 9 (9)
Subretinal fluid (Eye disorders) | 14 (17) | 14 (16)
Neovascular age-related macular degeneration (Eye disorders) | 8 (9) | 10 (12)
Influenza (Infections and infestations) | 9 (9) | 9 (9)
Nasopharyngitis (Infections and infestations) | 4 (5) | 12 (15)
Intraocular pressure increased (Investigations) | 7 (12) | 11 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02540954/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02540954/SAP_000.pdf